CLINICAL TRIAL: NCT02212288
Title: Antioxidant Signature in Adult Patients With Phenylketonuria (PKU) and Healthy Volunteers : Relationship With Metabolic Disturbances
Brief Title: Antioxidant Signature in Adult Patients With Phenylketonuria
Acronym: StressOX-PCU
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHAO14/FM-StressOX-PCU
Record Dates: First submitted 2014-07-28; First posted 2014-08-08 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: PKU; Hyperphenylalaninemia
MeSH Terms: conditions — Phenylketonurias | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PKU patients: Adult PKU patients;Blood samples;Urine sample only at inclusion
  Interventions: Other: Blood sample; Other: Urine sample
- Healthy controls: Adult Healthy controls;Blood samples;Urine samples only at inclusion
  Interventions: Other: Blood sample; Other: Urine sample

INTERVENTIONS:
Other: Blood sample — Blood samples are for metabolic and genetic and biological investigation
Other: Urine sample — Urine sample for biological investigation

SUMMARY:
To date, oxidative stress in PKU has been evaluated only with fragmented approaches.The aim of the present study is to investigate oxidative stress in PKU with more comprehensive methods.The relationship between oxidative stress and metabolic disturbances (hyperPhenylalaninemia) will also be studied.

DETAILED DESCRIPTION:
Analysis of oxidative stress

Oxidative metabolism is most likely disrupted leukocytes in the PCU thereof having DNA breaks correlated to blood Phe levels (22). Accessibility by patients, these cells are therefore interesting "tools" for analysis of oxidative stress in PKU.

-Hydrogen Peroxide intraleucocytaire We will isolate the leukocytes from heparinized samples to analyze intracellular H2O2 levels by flow cytometry after labeling with 5-(and 6)-chloromethyl-2 ', 7'-dicholorohydrofluorescein diacetate, acetyl ester (CM-H2DCFDA).

Anti-oxydogramme We will carry out an anti-oxydogramme which was the subject of a patent (Herault O & Vignon C "Method for Cancer Diagnosis" - Patent PCT / EP2011 / 073,757 filed Dec. 22, 2011) in the field of oncology. This is to achieve expression of an anti-oxidant genes in PKU profile compared with control subjects. This approach is based on three techniques: determining the level of expression of key antioxidants by RT-qPCR gene comparison with the expression of a housekeeping gene (GAPDH), ranked by their level of gene expression and comparison with the level of expression of the same genes in a reference pool RNA, used as internal calibrator. We will express these results through the RQ (relative quantification). The panel of antioxidant genes studied is the following: genes antioxidant enzyme systems not thiols: superoxide dismutase (SOD1, SOD2, SOD3) and catalase (CAT) or thiols: glutathione system (GPX, GPX1, GPX2, GPX3, GPX4, GPX5, GPX6, GPX7 GSR), the thioredoxin (TXN, TXN2) of peroxyredoxins (PRDX, PRDX2, PRDX4, PRDX5, PRDX6) and glutaredoxins (GLRX, GLRX2, GLRX3, GLRX5).

* Way NRF2 The NRF2 pathway H2O2 / being very classically activated when oxidative stress, we will quantify the expression of target genes NRF2 (HMOX, NQO1, GPX2). If they are overexpressed, the nuclear translocation of NRF2 be studied by confocal microscopy.
* DNA Breaks The breaks in DNA related to the oxidative stress in leukocytes are analyzed by flow cytometry (marking -H2AX) and electrophoretic migration of the fluorescent DNA (COMET assay).
* antioxidant vitamins and trace elements We will measure the plasma concentrations of vitamin A, C and E by a technique of liquid chromatography with UV detection. Furthermore, the activity of many enzymes is dependent antioxidant micronutrient, we doserons plasma concentrations of Se, Cu, Mn, and Zn.

Metabolic Balance

We realize chromatography plasma amino acids using the standard method of ion exchange chromatography with post-column derivation with ninhydrin. We will evaluate in particular the concentration of phenylalanine and tyrosine. We will focus on also other amino acids as described antioxidant potential (citrulline, taurine, histidine ...) We will evaluate by GC-MS organic acids commonly accumulated in the urine of PKU patients: dihydroxyphenylalanine, phenyllactate, phenylpyruvate, phenylacetate. Bioptérines concentrations and its derivatives will also be evaluated in HPLC with fluorescence detection.

ELIGIBILITY:
Inclusion Criteria:

* PKU patients over 18 years of age with phenylketonuria not treated with a phenylalanine-controlled diet.
* Affiliation to a social security scheme
* Reading and signing the informed consent
* Control subjects: all healthy subjects over 18 years of unfulfilled abnormal metabolism of whatever nature and associated symptoms

Exclusion Criteria:

* Pregnancy of patients and control subjects women (confirmed by a negative pregnancy test)
* Patients with diseases that may cause oxidative stress (neurodegenerative diseases, cancer)
* Patients treated with drugs known to cause oxidative stress
* Control subjects:controlled protein diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 PKU patients and 10 healthy controls with age and sex match
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of oxidative stress markers | First Day
  The main purpose of this preliminary study is to characterize oxidative stress in patients with PKU adults through a comprehensive approach involving the assessment of a wide combination of characteristic markers of oxidative stress and metabolic parameters that may be involved. In this context, we propose to establish an anti-oxidant signing in adult patients PCU using an innovative and comprehensive technical involving
  1. Quantification of intraleucocytaire hydrogen peroxide (Evaluated by flow cytometry and is expressed as relative fluorescence intensity between patients and the control group)
  2. Study of the expression of 24 genes involved in oxidative stress response (anti-oxydogramme)
  3. Comparison nuclear NRF2 translocation
  4. Comparison of DNA breaks
  5. Quantification of antioxidant vitamins and trace elements.(in difference from Normal values)

SECONDARY OUTCOMES:
Plasma concentrations of amino acids and organic acids concentration | First day
  Measurement of concentration of amino acids and organic acids concentration found in the 2 groups in comparison to normal values

CONTACTS AND LOCATIONS:
Overall Officials: François MAILLOT, MD-PhD, Study Director — University Hospital of TOURS, France
Locations (1):
- University Hospital of TOURS, Tours, I&L, France